CLINICAL TRIAL: NCT04327700
Title: A Phase II Study Of Intrabucally Administered Electromagnetic Fields and Regorafenib as Second-line Therapy For Patients With Advanced Hepatocellular Carcinoma.
Brief Title: Study Of Intrabucally Administered Electromagnetic Fields and Regorafenib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); THERABIONIC INC. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00064732; WFBCCC 55319 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Regorafenib and TheraBionic (Experimental): TheraBionic is a device that consists of battery-driven radiofrequency electromagnetic field generator. The metal mouth spoon antenna is placed on the anterior part of the tongue during treatment.
  Regorafenib is a 40 mg tablet administered orally.
  Interventions: Device: TheraBionic; Drug: Regorafenib

INTERVENTIONS:
Device: TheraBionic — Amplitude-modulated electromagnetic fields will be self-administered and given continuously to patients in three courses of 60-minute treatments per day, administered in the morning, at noon and in the evening at the patient's home, with the exception of the first 60-minute treatment, which will be delivered at the research site. Each 4 week treatment period will be considered a cycle of treatment.
  Other Names: Amplitude-modulated electromagnetic field device
Drug: Regorafenib — Patients will receive 160 mg regorafenib (four 40 mg tablets) orally once daily for the first 3 weeks of each 4-week cycle per approved prescribing information.
  Other Names: Stivarga

SUMMARY:
The primary goal of this study is to gather efficacy data concerning the progression-free survival rate with electromagnetic fields plus Regorafenib when compared to historical data with Regorafenib alone as a second-line therapy in patients with advanced hepatocellular carcinoma who have received any first line systemic therapy either standard of care Sorafenib or Lenvatinib or any experimental therapy. Patients who have received any treatment that includes either electromagnetic fields or Regorafenib will be excluded.

DETAILED DESCRIPTION:
Primary Objective: To estimate progression-free survival rates.

Secondary Objectives

* To obtain information concerning the feasibility of administration of the proposed treatment, including patient participation in trials using the proposed treatment.
* To evaluate safety and tolerability in this patient population.
* To evaluate the effect on levels of alpha-fetoprotein.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven hepatocellular carcinoma is locally advanced or metastatic. OR
* Patients without biopsy confirmation are also eligible if they meet the following:
* Radiologic diagnosis of hepatocellular carcinoma as per the American Association for the Study of Liver Diseases (AASLD) guidelines:
* liver cirrhosis AND
* a liver mass confirmed by blinded independent central review that shows arterial phase hyperenhancement on triphasic CT or MRI, AND EITHER:
* Is ≥20 mm with either non-peripheral portal washout or an enhancing capsule
* OR is 10-19 mm with non-peripheral portal venous washout AND an enhancing capsule.
* Patient must have been treated with at least one standard systemic treatment modality for advanced hepatocellular carcinoma such as sorafenib, lenvatanib, atezolizumab plus bevacizumab, or another approved or experimental systemic therapy prior to study entry.
* Measurable disease according to RECIST version 1.1 and mRECIST for hepatocellular carcinoma.
* At least one target lesion should not have previously received any local therapy, such as surgery, radiation therapy, hepatic arterial embolization, transarterial chemoembolization (TACE), hepatic arterial infusion, radio-frequency ablation, percutaneous ethanol injection or cryoablation, unless it has subsequently progressed by 20% or more according to RECIST version 1.1 and mRECIST for hepatocellular carcinoma.
* Patients with Child's Pugh A (at time of enrollment), with compensated cirrhosis, as defined by the parameters contained in the Child Pugh Calculator found in Appendix E.
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2
* Absence of medical or psychiatric contraindication which, in the opinion of the treating Investigator, would make the patient's participation in this trial inappropriate.
* Patient must not have curative treatment options, including surgery or radiofrequency ablation, available.
* Any extra-hepatic metastases, including treated central nervous system metastases but patients cannot have leptomeningeal disease.
* At least 2 weeks must have elapsed since administration of any anti-cancer treatment.
* Other anti-cancer treatments are not permitted during this study, including alternative medicine and herbal therapies.
* Patients must be 18+ years old and must be able to understand and sign an informed consent.
* Patient must agree to be followed up according to the study protocol.

Exclusion Criteria:

* Known leptomeningeal disease.
* Fibro lamellar hepatocellular carcinoma.
* Patients who had surgical resection of the disease and who do not have measurable disease.
* Patients with any of the following history within the 12 months prior to study drug administration: severe/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, including transient ischemic attack, or pulmonary embolism.
* Pregnant or breastfeeding women.
* Patients diagnosed with another type of cancer (excluding basal cell carcinoma) whose cancer diagnosed previously is not in remission.
* Patients receiving calcium channel blockers and any agent blocking L-type or T-type Voltage Gated Calcium Channels, e.g. amlodipoine, nifedipine, ethosuximide, etc. are not allowed in the study unless their medical treatment is modified to exclude calcium channel blockers prior to enrollment.
* Patients allergic or intolerant to Sorafenib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 12 weeks
  Progression-free survival will be estimated along with estimates of 95% confidence intervals for the treatment group. In addition, we will determine the proportion of patients who are progression free after 12 weeks (after 2nd 6-week visit) and compare this to the proportion of patients that were described as progression free in the RESORCE trial using a Simon's two stage design.

SECONDARY OUTCOMES:
Overall Survival | 6 months
  Kaplan Meier curves for patients survival and also estimate the percent of patients who are alive at 6 months and the corresponding 95% Clopper Pearson exact confidence intervals will be calculated.
Percentage of Participants with Disease Control | At 4 months and at 6 months from the date of enrollment
  Disease control is defined as the percentage of participants alive and have documented response status of complete response, partial response or stable disease according to the modified RECIST (mRECIST) for hepatocellular carcinoma using a 95% Clopper Pearson exact confidence interval. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of longest diameters of target lesions, without evidence of disease progression. Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Incidences of Adverse Events | Up to 30 days after treatment ends
  Type, incidence, severity of adverse events graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Adverse events will be described for each CTL type for this study using counts/percent's.
Comparison of Adverse Events (WFBCCC 55319 to RESORCE historical trial) | Up to 30 days after treatment ends
  Type, incidence, severity of adverse events graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
  Adverse events will be compared for each CTL type for the treatment group (WFBCCC 55319 study) and historical control (from the RESORCE trial), using the Fisher's exact test (two-sided) at level 0.05. These comparisons will be made to compare events of grade greater than or equal to 3 between each group.
Change in Alpha-fetoprotein Levels | 6 months
  Average alpha-fetoprotein level levels will be examined over time, and these changes in Alfa-fetoprotein rates after 6 months will be examined for each Response category (complete response/ partial response/ stable disease/ progressive disease) and tested using a 1-way ANOVA to see if the change in alpha-fetoprotein level differs by response category.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Paluri, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT04327700/ICF_000.pdf